CLINICAL TRIAL: NCT01529866
Title: A Prospective Randomized-controlled Study of the Integration Success Rate of an Implant System With a Novel Abutment Attachment in Cases Loaded Immediately
Brief Title: Study of the Integration Success of an Implant System With a Novel Abutment Attachment Design in Immediate Loading Cases
Acronym: Bridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3013
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: clinical study; edentulism; dental implants; Nanotite Certain Tapered implant; randomized; crestal bone level; immediate loading
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New abutment connection implant (Experimental): Implant with new abutment connection
  Interventions: Device: New Abutment Connection implant
- Nanotite Certain Tapered implant (Active Comparator): Nanotite Certain Tapered (standard abutment connection) implant
  Interventions: Device: Nanotite Certain Tapered implant

INTERVENTIONS:
Device: New Abutment Connection implant — New abutment connection implant
  Other Names: Osseotite Endosseous dental implant
  Arms: New abutment connection implant
Device: Nanotite Certain Tapered implant — Nanotite certain tapered (standard abutment connection) implant
  Other Names: Nanotite Endosseous dental implant
  Arms: Nanotite Certain Tapered implant

SUMMARY:
Integration success rates measured by lack of implant mobility and crestal bone regression measurement will be higher for the experimental implant design than for the control implants.

DETAILED DESCRIPTION:
In this study patients are randomized to receive either the experimental implant system or the control Nanotite Certain Tapered (standard abutment connection) and assessed for integration success measured by cumulative success rate in cases that are loaded immediately

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and older than 18 years of age
* patients needing at least one dental implant to treat partial edentulism
* patients physically able to tolerate surgical and restorative dental procedures
* patients agreeing to all protocol visits

Exclusion Criteria:

* patients with infection or severe inflammation at the intended treatment sites
* patients smoking greater than 10 cigarettes per day
* patients with uncontrolled diabetes mellitus
* patients with uncontrolled metabolic diseases
* patients who received radiation treatment to the head in the past 12 months
* patients needing bone grafting at the intended treatment sites
* patients known to be pregnant at screening visit
* patients with para-functional habits like bruxing and clenching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cumulative success rate | 2 years
  crestal bone regression (amount of bone loss measured) and equivalence in integration success (implant mobility)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Carvajal, DDS, Principal Investigator — University of Chile
Locations (1):
- Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No